CLINICAL TRIAL: NCT05210179
Title: Open-Label, Two Arms, Multi-Centered, Phase 2b Clinical Trial to Determine the Safety, Efficacy, and Immunogenicity of Booster Vaccination (TURKOVAC) Against SARS-CoV-2
Brief Title: Phase 2b Booster Vaccination (TURKOVAC) Against COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TSB-VAC-COV-TUR-RF2B.05
Record Dates: First submitted 2022-01-26; First posted 2022-01-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Sars-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 Vaccine; Booster; Efficacy; Immunogenicity; Safety
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: National, Open-Label, Two Arms, Multi-Centered, Phase 2b Clinical Trial to Determine the Safety, Efficacy, and Immunogenicity of Booster Vaccination (TURKOVAC) Against SARS-CoV-2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TURKOVAC-Koçak (Active Comparator): The dose of the TURKOVAC vaccine will be 3 μg/0.5 mL and will be administered by injection into the deltoid muscle.
  Interventions: Biological: TURKOVAC-Koçak
- TURKOVAC-Dollvet (Active Comparator): The dose of the TURKOVAC vaccine will be 3 μg/0.5 mL and will be administered by injection into the deltoid muscle.
  Interventions: Biological: TURKOVAC-Dollvet

INTERVENTIONS:
Biological: TURKOVAC-Dollvet — TURKOVAC-Dollvet vaccines produced by Dollvet Veterinary Vaccine Pharmaceutical Biological Substance Production Industry Co., Ltd.
  Arms: TURKOVAC-Dollvet
Biological: TURKOVAC-Koçak — TURKOVAC-Koçak vaccines produced by Koçak Farma Pharmaceutical and Chemical Industry Co., Ltd.
  Arms: TURKOVAC-Koçak

SUMMARY:
This study is open-label, two arms, multi-centered, phase 2b clinical trial to determine the efficacy, safety, and immunogenicity of booster vaccination (TURKOVAC) against Covid-19.

The primary aim of the study is to evaluate the efficacy of a booster dose of TURKOVAC vaccine administered to subjects who have passed at least 90 days and at most 240 days after the second dose of the first course of Comirnaty (Code name: BNT162b2) vaccine.

DETAILED DESCRIPTION:
This phase 2b study aims to determine the efficacy, safety, and immunogenicity of a booster dose of TURKOVAC vaccine administered to subjects who have passed at least 90 days and at most 240 days after the second dose of the first course of Comirnaty (Code name: BNT162b2) vaccine.

Efficacy will be evaluated by spike-specific antibody response and neutralizing antibody levels on days 0, 28 (all subjects), 48, 84 and 168 days (50% of subjects).

For the booster dose, subjects will be assigned open-label according to randomization (1:1) for 2 different arms. Comparing the efficacy, safety, and immunogenicity results of different series of TURKOVAC vaccines (TURKOVAC-Koçak and TURKOVAC-Dollvet) produced in different production facilities are the secondary objectives of the study.

The booster dose vaccine arms are as follows:

* TURKOVAC-Koçak
* TURKOVAC-Dollvet

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to give signed informed consent to participate in study,
2. Healthy male or female aged 18 - 59 years (including both groups),
3. Subjects who were vaccinated with Comirnaty (Code name: BNT162b2) for 2 doses and who had a minimum of 90 days and a maximum of 240 days after the second dose,
4. Subjects with a minimum of 28 days and a maximum of 42 days between 1st and 2nd dose of Comirnaty (Code name: BNT162b2) vaccines,
5. Female subjects of childbearing potential and male subjects of to have child potential who are willing to ensure that they or their partner use effective contraception continuously from 1 month before vaccination to 3 months after booster vaccination,
6. In the opinion of the investigator, subjects capable and willing to comply with all study requirements,
7. Subjects are willing to agree to abstain from donating blood during the study.

Exclusion Criteria:

1. Administration of any vaccine (registered or investigational) other than study intervention within 30 days before and after each study vaccine (one week for authorized seasonal flu vaccine or pneumococcal vaccine),
2. Known history of SARS-CoV-2 infection,
3. Pre-or planned use of another vaccine or product likely to affect the study (e.g. adenovirus vectored vaccines, any coronavirus vaccine),
4. Subjects who were pregnant at the time of enrollment or who plan to become pregnant within the first 3 months following vaccination and who are breastfeeding,
5. Subjects with fever (above 38°C) at the time of vaccination and/or up to 72 hours before (subjects may be screened again after acute condition has resolved),
6. Administration of immunoglobulins and/or any blood product within 3 months prior to vaccination,
7. Any confirmed or suspected immunosuppressive or immunodeficiency state; asplenia; recurrent severe infections and use of immunosuppressants (less than ≤14 days) in the last 6 months, excluding topical steroids or short-term oral steroids,
8. Possible history of allergic disease or reaction (e.g. to the active substance) by any component of the study vaccines,
9. Any history of anaphylaxis,
10. Current cancer diagnosis or treatment (excluding basal cell carcinoma of the skin and cervical carcinoma in situ),
11. History of bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture,
12. Continued use of anticoagulants such as coumarins and related anticoagulants (i.e. warfarin) or new oral anticoagulants (e.g. apixaban, rivaroxaban, dabigatran and edoxaban),
13. Cerebral venous sinus thrombosis, antiphospholipid syndrome, or a history of heparin-induced thrombocytopenia and thrombosis (HITT or HIT type 2),
14. Suspected or known current alcohol or drug addiction,
15. Any other significant disease, disorder or finding that could significantly increase the subject's risk for participation in the study, affect the subject's ability to participate in the study, or impair the interpretation of study data; severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, kidney disease, endocrine disorder, and neurological disease (mild/moderate well-controlled comorbidities are permitted),
16. History of active or previous autoimmune neurological disorders (e.g. multiple sclerosis, Guillain-Barre syndrome, transverse myelitis) (Bell's palsy will not be an exclusion criterion),
17. Subjects with severe renal impairment or liver failure,
18. Subjects who will undergo scheduled elective surgery during the study,
19. Subjects with a life expectancy of less than 6 months,
20. Subject who participated in another clinical trial study involving an investigational product in the past 12 weeks,
21. In case of clinical necessity, a COVID-19 PCR (polymerase chain reaction) test will be requested from the subjects, and subjects who are positive will be excluded from the study,
22. Known history of SARS-CoV-2 infection,
23. Acute respiratory disease (moderate or severe illness with or without fever). (Subjects may be screened again after acute condition has resolved),
24. Fever (greater than 37.8°C as measured by ear) (Subjects can be enrolled again after acute condition improves),
25. Insufficient level of Turkish to perform the informed consent, except where briefing by an independent witness can be provided and is available.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Neutralizing Antibodies | On days 0 and 28
  The change in the level of SARS-CoV2 Neutralizing Antibodies in the 28th day compared to the baseline
Pseudo-Neutralizing Antibodies | On days 0 and 28
  The change in the level of SARS-CoV2 Pseudo-Neutralizing Antibodies in the 28th day compared to the baseline
Anti-spike protein immunoglobulin G | On days 0 and 28
  The change in the level of SARS-CoV2 anti-spike protein immunoglobulin G in the 28th day compared to the baseline
T Cell Responses | On days 0 and 28
  The change in the level of T Cell Responses in the 28th day compared to the baseline

SECONDARY OUTCOMES:
Rates of subjects who have been found to be positive for COVID-19 | On day 0
  Rates of subjects who have been found to be positive for COVID-19 by RT-PCR (real time polymerase chain reaction) test after administration of TURKOVAC vaccine.
  (On day 0 and it will be repeated if the subject develops symptoms during the follow-up period)
Incidence of Adverse Reaction | Within 7 days of booster vaccination
  Incidence of adverse reactions within 7 days of vaccination in all subjects. (Within 7 days of booster vaccination)
Incidence of Serious Adverse Events (SAE) | Up to day 168 after booster vaccination
  Incidence of Serious Adverse Events (SAE) up to day 168 after vaccination in all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Bedia Dinç, Assoc. Prof., Principal Investigator — Faculty Member
Locations (9):
- Turkey (Türkiye) (9):
  - T.R. Ministry of Health Ankara City Hospital, Infectious Diseases and Clinical Microbiology Clinic, Ankara
  - University of Health Sciences, Antalya Training and Research Hospital, Family Medicine Clinic, Antalya
  - Abant İzzet Baysal University Izzet Baysal Training and Research Hospital, Bolu
  - İstanbul University Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Department of Internal Medicine - Department of Infectious Diseases and Clinical Microbiology, Istanbul
  - T.R. Ministry of Health Başakşehir Çam ve Sakura City Hospital, Clinical Microbiology Clinic, Istanbul
  - T.R. Ministry of Health Istanbul Provincial Health Directorate Prof. Dr. Cemil Taşçıoğlu City Hospital, Infectious Diseases and Clinical Microbiology Clinic, Istanbul
  - T.R. Ministry of Health İzmir Provincial Health Directorate İzmir Health Sciences University Tepecik Training and Research Hospital, Infectious Diseases, Izmir
  - T.R. Ministry of Health Kayseri City Training and Research Hospital, Infectious Diseases and Clinical Microbiology Department, Kayseri
  - University of Health Sciences, Derince Training and Research Hospital, Department of Infectious Diseases and Clinical Microbiology, Kocaeli